CLINICAL TRIAL: NCT04614805
Title: Mobilizing Clinical Leadership to Achieve Timely Reperfusion in Acute ST-segment Elevation Myocardial Infarction
Brief Title: Timely Reperfusion in Acute ST-segment Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Kristian Bartnes, Director of Division of Cardiothoracic and Respiratory Medicine, University Hospital of North Norway
Other Study IDs: iTide
Record Dates: First submitted 2020-10-18; First posted 2020-11-04 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mobilizing clinical leaders — Clinical leaders and clinical personnel will regularly receive feedback regarding performance of their own hospital as well as other providers in the regional health trust of North Norway.

SUMMARY:
The aim of the study is to monitor outcomes, especially time to reperfusion, in ST-elevation acute myocardial infarction patients.

DETAILED DESCRIPTION:
In the regional health trust of North Norway, time to reperfusion in acute ST-elevation myocardial infarction is below the national average and below recommendations. The aim of this study is to monitor outcomes, especially time to reperfusion, in ST-elevation acute myocardial infarction patients. The study period is supposedly lasting for approximately 4 months, the time estimated to observe the clinical course of 100 patients. Before and during the study period, clinical leaders are encouraged to improve guideline adherence and to closely monitor the results of their own and collaborating institutions.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with acute myocardial infarction with ST-elevations within our regional health trust during Nov 1st and for approx 4 months, and with an indication for reperfusion therapy (thrombolysis and/pr PCI)

Exclusion Criteria:

* Reperfusion therapy not indicated or contraindicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with STEMI in our regional health trust during the study period who has an indication for immediate reperfusion therapy
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Time to reperfusion | This parameter will be recorded within 1 week after patient inclusion
  Interval between 1st medical contact and opening of the infarction-related coronary artery.

SECONDARY OUTCOMES:
Ejection fraction at discharge | This parameter will be recorded up to 6 months after patient inclusion
  Systolic function of the left ventricle
Survival | This parameter will be collected from patient's records during Nov -20 till Aug -21.
  Survival after 30 days from incident

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital North Norway, Tromsø, Troms Og Finnmark, Norway

IPD SHARING:
Plan to Share IPD: Undecided
so far no plans for such sharing.

REFERENCES:
- [Derived] Bartnes K, Albrigtsen H, Iversen JM, Brovold H, Moller NH, Wembstad B, Arstad F, Kristensen AH, Cortis J, Olsen SJ, Nygaard SNS, Kindler SG, Moe O, Hansen C, Mannsverk JT. The Barriers to Rapid Reperfusion in Acute ST-Elevation Myocardial Infarction. Cardiol Ther. 2022 Dec;11(4):559-574. doi: 10.1007/s40119-022-00281-7. Epub 2022 Oct 6. PMID 36203049